CLINICAL TRIAL: NCT02885532
Title: The University of California, San Diego Brief Assessment of Capacity to Consent Instrument in Acutely Intoxicated Emergency Department Patients
Brief Title: Capacity to Consent in Acutely Intoxicated Emergency Department Patients
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 15-3949
Record Dates: First submitted 2016-08-24; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Informed Consent
Keywords: alcohol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: University of California, San Diego Brief Assessment of Capacity to Consent Tool — Non-pregnant, English speaking patients older than 18 with evidence of acute alcohol intoxication were considered eligible for participation. Patients were asked to complete the 10 question tool on arrival to the emergency department. Patie

SUMMARY:
The ability to meaningfully consent intoxicated and chemically dependent patients for research has inhibited medical advances in this vulnerable population. A recent pilot supported use of the University of California, San Diego Brief Assessment of Capacity to Consent tool to assess the capacity of intoxicated emergency department patients to participate in research. The objective is to determine the number of intoxicated emergency department patients who could correctly complete the questionnaire, and evaluate alcohol concentration, sedation and ability to recall participation upon sobriety.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, intoxicated with alcohol

Exclusion Criteria:

* intoxication was due to a substance other than ethanol (negative breath alcohol concentration), refusal to participate, excessive agitation, or if the treating physician deemed the patient medically or psychologically unstable. Patients were also excluded if they had previously been enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-pregnant, English speaking patients aged 18 years or older with clinical evidence of acute alcohol intoxication as the predominant etiology of mental status changes were eligible.
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The number of intoxicated emergency department patients who could correctly complete the questionnaire | Immediately

SECONDARY OUTCOMES:
Alcohol concentration (breath or serum) | Immediately
Degree of sedation | Immediately
  Observer's Assessment of Alertness/Sedation scale (OAA/S) score
Recall of participation | Between 2 and 12 hours after initial enrollment, depending on the time clinical sobriety achived

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCormack RP, Gallagher T, Goldfrank LR, Caplan AL. Including frequent emergency department users with severe alcohol use disorders in research: assessing capacity. Ann Emerg Med. 2015 Feb;65(2):172-7.e1. doi: 10.1016/j.annemergmed.2014.09.027. Epub 2014 Oct 23. PMID 25447556